CLINICAL TRIAL: NCT02068664
Title: An Assessment of the Prevalence of Spatial Neglect in Stroke Survivors With Aphasia With Option of Prism Adaptation Treatment (PAT) Protocol
Brief Title: An Assessment of the Prevalence of Spatial Neglect in Stroke Survivors With Aphasia
Status: Completed | Type: Observational
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: R-802-13
Record Dates: First submitted 2014-02-12; First posted 2014-02-21 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Spatial Neglect; Aphasia; Stroke
Keywords: spatial neglect; aphasia
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational: prism adaptation treatment
  Interventions: Behavioral: prism adaptation treatment

INTERVENTIONS:
Behavioral: prism adaptation treatment — Prism goggles shift the image one sees toward the left (because the thicker portion of the glass lens is on the right). This will change the perception of where the image is in space, causing the person to adapt. The after-effects of the treatment is what is important. It has been shown to make it easier for people to move in the right space (if have right neglect) or improves ability to complete other functional tasks.

SUMMARY:
The purpose of this study is to determine if stroke survivors with aphasia have spatial neglect (Phase 1). If they are determined to have the condition Phase 2 will be offered: which is prism adaptation treatment. This is a pilot study that will be performed with 4-5 subjects.

DETAILED DESCRIPTION:
Spatial neglect is a disorder that may occur after a brain injury such as stroke. Spatial neglect may affect stroke recovery. One example of this heterogeneous condition: Individuals with spatial neglect often pay more attention to one side of what they are looking at, even though they have no difficulty seeing. The study investigators would like to screen stroke survivors with aphasia because they may also have spatial neglect (right neglect after left hemisphere stroke), which is said by the literature to occur in 25% of cases. If it is identified, a treatment approach will be offered, to attempt to remediate the condition using prism goggles, following a prism treatment protocol based on previous studies.

ELIGIBILITY:
Inclusion Criteria:

* A stroke survivor with aphasia who is a member at the Adler Aphasia Center

Exclusion Criteria:

* Has a history of brain tumor, head injury with loss of consciousness, dementia, alzheimers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors with aphasia and spatial neglect
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Kessler Foundation Neglect Assessment Process | 2 weeks
  a performance based and behavioral measure for spatial neglect that utilizes and standardizes the administration of the Catherine Bergego Scale (CBS)

SECONDARY OUTCOMES:
Behavior Inattention Test | 2 weeks
  Conventional subtest, a set of paper and pencil test for spatial neglect
Barthel Index | 2 weeks
  A functional independence assessment of daily tasks
University of Alabama at Birmingham (UAB) Life Space assessment | 2 weeks
  a self graded assessment on community mobility and participation

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Hreha, OT, Principal Investigator — Kessler Foundation/Kessler Institute for Rehabilitation; A.M. Barrett, M.D., Principal Investigator — Kessler Foundation
Locations (1):
- Adler Aphasia Center, Maywood, New Jersey, United States

REFERENCES:
- See also: Kessler Foundation — http://kesslerfoundation.org